CLINICAL TRIAL: NCT05265052
Title: A Multicenter, Randomized, Phase IIa/IIb Clinical Trial of 3D1002 Combined With Oxycodone Hydrochloride Sustained-release Tablets in the Treatment of Patients With Moderate to Severe Cancer Pain
Brief Title: 3D1002 in Combination With Oxycodone Hydrochloride Sustained-release Tablets in Patients With Moderate to Severe Cancer Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 3D Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D1002-CN-001
Record Dates: First submitted 2022-01-24; First posted 2022-03-03 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cancer Pain
Keywords: Cancer pain
MeSH Terms: conditions — Cancer Pain | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Both phase IIa and IIb are randomized, parallel controlled studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 3D1002 50 mg group (Phase IIa) (Experimental): 3D1002 is given 50 mg twice a day for 2 weeks.
  Interventions: Drug: 3D1002 (50 mg)(Phase IIa)
- 3D1002 100 mg group (Phase IIa) (Experimental): 3D1002 is given 100 mg twice a day for 2 weeks.
  Interventions: Drug: 3D1002 (100 mg)(Phase IIa)
- 3D1002 150 mg group (Phase IIa) (Experimental): 3D1002 is given 150 mg twice a day for 2 weeks.
  Interventions: Drug: 3D1002 (150 mg)(Phase IIa)
- 3D1002 monotherapy group (Phase IIb) (Experimental): 3D1002 at recommended dose plus mimic OxyContin tables, will be given twice a day for 2 weeks.
  Interventions: Drug: 3D1002 monotherapy (Phase IIb)
- OxyContin monotherapy group (Phase IIb) (Experimental): OxyContin initiating at 10mg per dose plus mimic 3D1002 tablets, will be given twice a day for 2 weeks.
  Interventions: Drug: OxyContin monotherapy (Phase IIb)
- 3D1002 + OxyContin group (Phase IIb) (Experimental): 3D1002 at recommended dose plus OxyContin initiating at 10 mg per dose, will be given twice a day for 2 weeks.
  Interventions: Drug: 3D1002 + OxyContin (Phase IIb)

INTERVENTIONS:
Drug: 3D1002 (50 mg)(Phase IIa) — 1 tablet of 3D1002 per oral dose
  Arms: 3D1002 50 mg group (Phase IIa)
Drug: 3D1002 (100 mg)(Phase IIa) — 2 tablets of 3D1002 per oral dose
  Arms: 3D1002 100 mg group (Phase IIa)
Drug: 3D1002 (150 mg)(Phase IIa) — 3 tablets of 3D1002 per oral dose
  Arms: 3D1002 150 mg group (Phase IIa)
Drug: 3D1002 monotherapy (Phase IIb) — 3D1002 is administered at recommended dose with mimic OxyContin tablets.
  Arms: 3D1002 monotherapy group (Phase IIb)
Drug: OxyContin monotherapy (Phase IIb) — OxyContin is administered at an initial dose of 10 mg per dose with mimic 3D1002 tablets.
  Arms: OxyContin monotherapy group (Phase IIb)
Drug: 3D1002 + OxyContin (Phase IIb) — 3D1002 is administered at recommended dose, and OxyContin is administered at an initial dose of 10 mg per dose.
  Arms: 3D1002 + OxyContin group (Phase IIb)

SUMMARY:
This study aims to evaluate the safety and efficacy of 3D1002 alone or in combination with oxycodone hydrochloride sustained-release tablets (OxyContin) for the management of moderate or severe cancer pain.

DETAILED DESCRIPTION:
The investigational product in this study, 3D1002, is a selective antagonist of prostaglandin E2 receptor subtype 4 (EP4). The study is composed of two stages. Phase IIa stage is to assess the safety and efficacy of 3D1002 administered at doses of 50, 100 or 150 mg every 12 hour (q12h) for patients with moderate to severe cancer pain, and to determine the optimal recommended dose for further studies. Phase IIb stage is to evaluate the difference in the efficacy and safety of 3D1002 combined with OxyContin and OxyContin alone in treatment of patients with moderate to severe cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign the informed consent in person prior to beginning any screening procedure.
2. Age ≥18, both male and female.
3. Subjects with a malignant tumor confirmed by histopathology or cytology.
4. Weight ≥40 kg at screening period.
5. Subjects have relatively stable cancer pain and require continuous analgesic medications (estimated treatment duration ≥2 weeks), as assessed by the investigator.
6. Estimated life expectancy ≥3 months.
7. Subjects are willing to not use any analgesic other than those specified in the study during the study treatment period.
8. ECOG PS score is 0-3.
9. Have adequate organ and bone marrow function.
10. The mean NRS scores per day during the washout period are ≥4.

Exclusion Criteria:

1. Known allergy to any of the active ingredients or excipients of the study drug, or have a history of allergy to other opioids or non-steroidal anti-inflammatory drugs (NSAIDs) and their related ingredients.
2. Have a persistent pain resulted from other medical conditions or unknown causes.
3. Subjects presenting with emergency symptoms such as intestinal obstruction/perforation, spinal cord compression, epidural metastasis, or fracture.
4. Subjects with known active/symptomatic central nervous system metastasis and/or cancerous meningitis.
5. Subjects plan to be treated with >10 mg/ day of prednisone or equivalent systemic corticosteroid during the study period.
6. Have a history of gastrointestinal bleeding or perforation.
7. Have a positive result of fecal occult blood test during screening period.
8. Have a history of serious cardiovascular diseases.
9. Have a history of an acute ischemic or hemorrhagic stroke within 6 months prior to screening.
10. Have a history of significant psychiatric disorders, such as schizophrenia and depression.
11. Subjects plan to receive radiotherapy, surgery, or a new regimen of systemic antitumor agents during the study treatment period (D1-D15).
12. Subjects have a history of alcohol abuse or drug abuse including opioids.
13. Subjects have significant opioid contraindications.
14. Pregnant or lactating women.
15. Subjects with other diseases that affect the oral administration or absorption of drugs.
16. Subjects are currently participating in another clinical study.
17. Other conditions deemed by the investigator to be inappropriate for participation in this study, such as poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sum of pain intensity difference in the Numeric Rating Scale (NRS) within 14 days after the first study drug treatment (SPID14) | 1 to 14 days after receiving study treatment
  ①Average pain intensity is calculated daily for the past 24 hours using the NRS (0 = No pain, 10 = Worst pain imaginable). ②PID (pain intensity difference): Baseline pain intensity score (for the day prior to the day of randomization) minus pain intensity score at each given day.③SPID: the sum of the pain intensity difference generated daily from day 1 to the designated day.

SECONDARY OUTCOMES:
Proportion of subjects who achieve effective pain control | 1 to 14 days after receiving study treatment
  Effective pain control: mean NRS score within 0-3 points and episode of breakthrough pain ≤ 2 times in 24 hours
Time to achieve effective pain control | 1 to 14 days after receiving study treatment
Time-specific pain intensity difference（PID） | 1 to 14 days after receiving study treatment
Sum of pain intensity difference (SPID) in the NRS within 3,5 and 7 days post-treatment | from day 1 to 3, 5 and 7 after receiving study treatment, respectively
Time-specific subject self-rated pain relief based on Brief Pain Inventory Short Form (BPI-SF) Questionnaire Item 8 | 1 to 14 days after receiving study treatment
  The pain relief is assessed daily for the past 24 hours based on the percentage of relief from baseline, ranging from 0 (no relief) to 100% (complete relief).
Sum of subject self-rated pain relief based on BPI-SF Questionnaire Item 8 within 3,5,7 and 14 days post-treatment | from day 1 to 3, 5, 7 and 14 after receiving study treatment, respectively
Proportion of subjects with pain response over 7 and 14 days after treatment | 1 to 14 days after receiving study treatment
  Pain response: at least 30% and 50% decrease in pain intensity NRS score from baseline.
Time to pain response | 1 to 14 days after receiving study treatment
The number of breakthrough pain episodes and rescue dose of immediate-release oxycodone over 7 and 14 days after treatment; | 1 to 14 days after receiving study treatment
Time-specific oxycodone dose, including immediate-release oxycodone capsules and sustained-release oxycodone tablets (the latter is only applicable for phaseⅡb) | 1 to 14 days after receiving study treatment
Total dose of oxycodone over 3, 7, and 14 days post-treatment | 1 to 14 days after receiving study treatment
Evaluation of the subjects' quality of life over 7 and 14 days after treatment by using of European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 V3.0) (for phase Ⅱb only) | 1 to 14 days after receiving study treatment
  EORTC QLQ-C30 comprises 30 items, including five functioning scales, a global quality of life (QoL) scale, three symptom scales and six single items. For the functioning and the global QoL scales, a higher score denotes better health. For the symptom scales and single-item scales, a higher score indicates more symptom burden.
Patient's global impression of change (PGI-C) over 7 and 14 days after treatment (for phase IIb only) | 1 to 14 days after receiving study treatment
  PGI-C is a participant rated instrument to measure participant's change in overall status of general condition including pain on a 7-point scale, with 1 being "very much improved" and 7 being "very much worse".
Frequency and severity of adverse events during treatment | 1 to 14 days after receiving study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No